CLINICAL TRIAL: NCT01462097
Title: Randomized Trial of Aerobic Exercise Training on Cognitive and Physical Function in Chronic Kidney Disease
Brief Title: Exercise Trial in Chronic Kidney Disease
Acronym: AWARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stephen Seliger, Associate Professor of Medicine at University of Maryland, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HP-00045276; 1R01DK090401-01A1 (NIH)
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Exercise; Aerobic capacity; Learning and memory; Executive function; Endothelial function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic exercise (Experimental): 12 months of treadmill walking and strength training exercise. Exercise is gradually progressed in walking speed and time on the treadmill based on the individual's tolerance, abilities, and safety. For months 1-6 exercise will take place 3 times per week at the research center. For months 6-12 exercise will take place 2 times per week at the center and 1 time per week at home.
  Interventions: Behavioral: Aerobic exercise training
- Health Education (Active Comparator): 12 months of Health education sessions which will cover topics important to older adults (safe travel, age-appropriate preventative screenings, resources for reliable health information, and topics relevant to chronic kidney disease). For months 1-6 classes will take place 1 time per week. For months 6-12 classes will take place 1 time per month.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Aerobic exercise training — 12 months of aerobic exercise
  Arms: Aerobic exercise
Behavioral: Health Education — 12 months of health education sessions
  Arms: Health Education

SUMMARY:
Chronic Kidney Disease (CKD) is exceedingly common in older adults, in whom it is associated with impairment in cognition and physical function. The purpose of this study is to test the effects of 12 months of aerobic and resistance exercise training compared to health education on cognitive and physical performance in 120 older adults with CKD not requiring dialysis. The results of this study will be essential for demonstrating the effectiveness of exercise in improving function and ultimately preventing disability in this high-risk population of older adults.

DETAILED DESCRIPTION:
This is a parallel-group randomized controlled trial comparing 12 months of aerobic and resistance exercise training vs. health education (attention control) on neurocognitive and physical performance among community-dwelling older adults (age >55) and CKD stage 3b and 4. Co-primary outcomes are change in physical performance (including aerobic capacity and submaximal walking) and neurocogntive performance (including executive functions).

Outcome measures will be assessed at baseline and after 6- and 12 months. Exercise training will occur thrice weekly at a dedicated research exercise center and will be supervised by exercise specialists.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3-4 Chronic kidney disease (estimated Glomerular Filtration Rate 15-45)
* Age 60 to 85
* English Speaking

Exclusion Criteria:

* Dementia or cognitive impairment
* Renal transplant
* New York Heart Association class 3-4 heart failure
* Severe Chronic Lung Disease
* Unstable angina or coronary revascularization within the last 3 months
* Orthopedic problems that would preclude aerobic exercise training
* Known, untreated infection
* Disabling arthritis
* Uncontrolled arrhythmia
* More than 14 alcoholic drinks per week

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-03; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baltimore VA Medical Center / University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Liu CK, Miao S, Giffuni J, Katzel LI, Fielding RA, Seliger SL, Weiner DE. Geriatric Syndromes and Health-Related Quality of Life in Older Adults with Chronic Kidney Disease. Kidney360. 2023 Apr 1;4(4):e457-e465. doi: 10.34067/KID.0000000000000078. Epub 2023 Feb 14. PMID 36790849
- [Derived] Weiner DE, Liu CK, Miao S, Fielding R, Katzel LI, Giffuni J, Well A, Seliger SL. Effect of Long-term Exercise Training on Physical Performance and Cardiorespiratory Function in Adults With CKD: A Randomized Controlled Trial. Am J Kidney Dis. 2023 Jan;81(1):59-66. doi: 10.1053/j.ajkd.2022.06.008. Epub 2022 Aug 6. PMID 35944747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2012 through June 2016 recruited from the University of Maryland Medical Center, VA Maryland Healthcare System, Tufts Medical Center, and Partners Healthcare.
Period: Overall Study
Arm/Group | Aerobic Exercise | Health Education
Started | 49 | 50
6 Month | 35 | 37
Completed | 30 | 38
Not Completed | 19 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | Health Education | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (7.7) | 68.1 (8.8) | 68.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 34 | 40 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 27 | 34 | 61
  Caucasian | 18 | 13 | 31
  Other | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 34.1 (9.5) | 32.6 (11.4) | 33.3 (10.5)
Hemoglobin (g/dl) [Mean (Standard Deviation); unit: g/dL] | 12.5 (1.6) | 12.3 (1.7) | 12.4 (1.6)
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 30.3 (7.2) | 31.8 (5.8) | 31.1 (6.5)
Self-reported Moderate-vigorous physical activity [Mean (Standard Deviation); unit: minutes/week] | 72 (126) | 90 (174) | 78 (150)
Coronary Artery Disease [Count of Participants; unit: Participants] | 16 | 13 | 29
Diabetes [Count of Participants; unit: Participants] | 30 | 28 | 58
Hypertension [Count of Participants; unit: Participants] | 44 | 48 | 92
Heart Failure [Count of Participants; unit: Participants] | 6 | 4 | 10
Peripheral vascular disease [Count of Participants; unit: Participants] | 3 | 6 | 9
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] | 5 | 8 | 13
Study Site [Count of Participants; unit: Participants]
  Tufts | 21 | 22 | 43
  Univ Maryland | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Aerobic Capacity
Description: VO2peak, measured by Graded Exercise Treadmill Test (GXT) with a modified Balke protocol - higher indicates better aerobic capacity
Time Frame: Baseline, 6 months, 12 months
Population: Participants with complete V02peak at >=1 time point
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Aerobic Exercise | Health Education
Number analyzed (Participants) | 48 | 50
ml/kg/min
  Baseline | 17.1 (5.3) | 16.8 (5.6)
  6 months: number analyzed (Participants) | 32 | 32
  6 months | 17.9 (5.5) | 15.9 (7.0)
  12 Months: number analyzed (Participants) | 25 | 37
  12 Months | 18.7 (5.2) | 17.2 (6.4)

2. Primary Outcome: Change in 6 Minute Walk
Description: Distance walked in 6 minutes - greater distance represents higher function
Time Frame: Baseline, 6 months, 12 months
Population: Total # with at least one measurement
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Aerobic Exercise | Health Education
Number analyzed (Participants) | 49 | 50
Feet
  Baseline | 1298 (323) | 1251 (394)
  6 months: number analyzed (Participants) | 35 | 37
  6 months | 1649 (620) | 1247 (454)
  12 months: number analyzed (Participants) | 29 | 37
  12 months | 1453 (368) | 1284 (462)

3. Secondary Outcome: Change in Physical Function
Description: Timed Up and Go Test
Time Frame: Baseline, 6 months, 12 months
Population: # of participants with complete measures
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Aerobic Exercise | Health Education
Number analyzed (Participants) | 49 | 49
Seconds
  Baseline | 8.2 (2.4) | 8.6 (2.7)
  6 months: number analyzed (Participants) | 34 | 33
  6 months | 8.0 (2.6) | 9.3 (3.6)
  12 months: number analyzed (Participants) | 29 | 36
  12 months | 8.3 (29) | 9.0 (2.9)

4. Secondary Outcome: Number With Short Physical Performance Battery (SPPB) Score <10 (Out of 12 Maximum)
Description: Short Physical Performance Battery is a test of lower extremity function designed to be administered in older adults, consisting of three components: 1) usual gait speed over a 4-meter course; 2) five repeated chair stands; 3) standing balance battery. Each component is scored 0-4, with higher scores indicating better function, and the total scores of each component are summed (range, 0-12).
Time Frame: Baseline, 6 months, 12 months
Population: # of participants with complete measures
Measure: Count of Participants; unit: Participants
Arm/Group | Aerobic Exercise | Health Education
Number analyzed (Participants) | 49 | 50
Participants
  Baseline | 19 | 19
  6 months: number analyzed (Participants) | 26 | 37
  6 months | 9 | 15
  12 months: number analyzed (Participants) | 29 | 36
  12 months | 9 | 16

ADVERSE EVENTS:
Time Frame: 12 months or until loss to follow-up or withdrawal.
Arm/Group | Aerobic Exercise | Health Education
All-Cause Mortality (participants affected / at risk) | 1/49 | 2/50
Serious Adverse Events (participants affected / at risk) | 21/49 | 34/50
Other Adverse Events (participants affected / at risk) | 30/49 | 31/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise (N=49) | Health Education (N=50)
All SAEs (General disorders) | 21 (21) | 34 (34) — SAEs were not categorized by organ system or type
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise (N=49) | Health Education (N=50)
All AEs (General disorders) | 30 (66) | 31 (79) — Adverse Events were not categorized by organ system or type

LIMITATIONS AND CAVEATS:
1. Study did not meet accrual target
2. Drop-out and loss to follow-up greater than expected, often to due to intercurrent medical events .
3. Moderately greater loss to follow-up in group randomized to exercise training
4. Lack of blinding of outcome assessors
5. Study not designed to have sufficient power to detect effects on secondary outcomes including kidney function.
6. No adjustment for multiple comparisons - risk of type 1 error may be greater than estimated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT01462097/Prot_000.pdf